CLINICAL TRIAL: NCT05612880
Title: Assessing Physical Function Following Androgen Receptor Signaling Inhibitor Treatment for Metastatic Prostate Cancer
Brief Title: Physical Function During ARSI Treatment
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2214
Record Dates: First submitted 2022-10-19; First posted 2022-11-10 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Advanced Prostate Carcinoma
Keywords: androgen deprivation therapy; ARSI; physical function
MeSH Terms: interventions — abiraterone; enzalutamide; darolutamide; apalutamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-intervention controls: Men with advanced prostate cancer initiating androgen receptor signaling inhibitor treatment.
  Interventions: Drug: androgen receptor signaling inhibitors

INTERVENTIONS:
Drug: androgen receptor signaling inhibitors — Prior to or within 8 weeks of ARSI initiation, men with advanced prostate cancer will perform baseline testing, with follow ups at 12 and 24 weeks
  Other Names: abiraterone; enzalutamide; darolutamide; apalutamide

SUMMARY:
This single arm observational pilot study aims to determine the longitudinal effects of androgen receptor signaling inhibitors (ARSI) in men with advanced prostate cancer. The primary outcome for this trial is physical function, which will be evaluated at baseline, 12 and 24 weeks. Secondary outcomes including body composition, muscle function, balance, arterial stiffness and patient reported outcomes.

DETAILED DESCRIPTION:
The purpose of this pilot trial is to obtain objective measurements of physical function in men with metastatic prostate cancer (mPC) initiating ARSI treatment at baseline, 12, and 24 weeks later. Grip strength, muscular power, body composition, balance, arterial stiffness, along with QoL, fatigue, anxiety, and depression will also be measured. Finally, the potential associations in primary and secondary outcomes by the type of ARSI, stage of mPC, and physical activity levels will be explored.

With more men requiring ARSI treatment for metastatic castrate resistant prostate cancer (mCRPC), as well as being an efficacious option earlier in metastatic castrate sensitive prostate cancer (mCSPC), accurate estimates of declines from ARSI initiation are required to determine the true effects. Utilizing novel assessments in mPC like muscular power tests will provide insight into potentially more relevant assessments and outcomes to intervene on. The data from this pilot study will also determine effect sizes to adequately power future studies.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Subjects is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.
* Age ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Diagnosis of metastatic disease from prostate cancer, or recurrent disease following definitive local therapy of prostate cancer, as assessed by their clinician
* Initiation of an ARSI (e.g., abiraterone, enzalutamide, apalutamide, or darolutamide) for mPC with concurrent androgen deprivation therapy (ADT).
* Availability to begin baseline testing within 8 weeks of ARSI treatment initiation.
* Physician clearance to perform physical assessments.
* Ability to speak and read English.

Exclusion Criteria:

* Prior ARSI treatment
* Current chemotherapy
* History of bone fractures or musculoskeletal injuries
* Neurological conditions that affect balance and/or muscle strength
* Intention to leave the region prior to completion of study
* Dementia, altered mental status or any psychiatric condition prohibiting the understanding or rendering of informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with metastatic prostate cancer, or recurrent disease following definitive local treatment, on androgen deprivation therapy, who are initiating treatment with androgen receptor signaling inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Physical function: 400m Walk | Baseline
  The time to walk 400m (in sec) will be performed as an indicator of walking endurance. A lower total time (and therefore higher gait speed) indicates greater cardiorespiratory capacity.
Physical function: 400m Walk | 12 weeks
  The time to walk 400m (in sec) will be performed as an indicator of walking endurance. A lower total time (and therefore higher gait speed) indicates greater cardiorespiratory capacity.
Physical function: 400m Walk | 24 weeks
  The time to walk 400m (in sec) will be performed as an indicator of walking endurance. A lower total time (and therefore higher gait speed) indicates greater cardiorespiratory capacity.
Physical function: Timed Up and Go | Baseline
  The time to complete (in sec) the 2.44m (8 ft) timed up and go test will be performed as an indicator of agility, balance, and physical function. A lower total time is indicative of greater performance.
Physical function: Timed Up and Go | 12 weeks
  The time to complete (in sec) the 2.44m (8 ft) timed up and go test will be performed as an indicator of agility, balance, and physical function. A lower total time is indicative of greater performance.
Physical function: Timed Up and Go | 24 weeks
  The time to complete (in sec) the 2.44m (8 ft) timed up and go test will be performed as an indicator of agility, balance, and physical function. A lower total time is indicative of greater performance.
Physical function: Short physical performance battery | Baseline
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability. Clinically meaningful changes are 0.3-1.0 points.
Physical function: Short physical performance battery | 12 weeks
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability. Clinically meaningful changes are 0.3-1.0 points.
Physical function: Short physical performance battery | 24weeks
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability. Clinically meaningful changes are 0.3-1.0 points.

SECONDARY OUTCOMES:
Body composition: lean mass | Baseline
  To report total body lean mass using dual-energy x-ray absorptiometry (DXA).
Body composition: lean mass | 12 weeks
  To report total body lean mass using dual-energy x-ray absorptiometry (DXA).
Body composition: lean mass | 24 weeks
  To report total body lean mass using dual-energy x-ray absorptiometry (DXA).
Body composition: fat mass | Baseline
  To report total body fat mass using dual-energy x-ray absorptiometry (DXA).
Body composition: fat mass | 12 weeks
  To report total body fat mass using dual-energy x-ray absorptiometry (DXA).
Body composition: fat mass | 24 weeks
  To report total body fat mass using dual-energy x-ray absorptiometry (DXA).
Body composition: bone mass | Baseline
  To report total body bone mass using dual-energy x-ray absorptiometry (DXA).
Body composition: bone mass | 12 weeks
  To report total body bone mass using dual-energy x-ray absorptiometry (DXA).
Body composition: bone mass | 24weeks
  To report total body bone mass using dual-energy x-ray absorptiometry (DXA).
Body composition: thigh muscle cross-sectional area | Baseline
  Muscle size will be analyzed using ultrasound of the vastus lateralis of the dominant leg. Higher muscle mass and quality are associated with greater muscle strength, physical function, QoL, and mortality.
Body composition: thigh muscle cross-sectional area | 12 weeks
  Muscle size will be analyzed using ultrasound of the vastus lateralis of the dominant leg. Higher muscle mass and quality are associated with greater muscle strength, physical function, QoL, and mortality.
Body composition: thigh muscle cross-sectional area | 24 weeks
  Muscle size will be analyzed using ultrasound of the vastus lateralis of the dominant leg. Higher muscle mass and quality are associated with greater muscle strength, physical function, QoL, and mortality.
Body composition: thigh muscle quality | Baseline
  Muscle architecture will be analyzed using ultrasound of the vastus lateralis of the dominant leg. Higher muscle mass and quality are associated with greater muscle strength, physical function, QoL, and mortality. Muscle quality is reported in arbitrary units, where a lower value indicates a higher/better muscle quality.
Body composition: thigh muscle quality | 12 weeks
  Muscle architecture will be analyzed using ultrasound of the vastus lateralis of the dominant leg. Higher muscle mass and quality are associated with greater muscle strength, physical function, QoL, and mortality. Muscle quality is reported in arbitrary units, where a lower value indicates a higher/better muscle quality.
Body composition: thigh muscle quality | 24 weeks
  Muscle architecture will be analyzed using ultrasound of the vastus lateralis of the dominant leg. Higher muscle mass and quality are associated with greater muscle strength, physical function, QoL, and mortality. Muscle quality is reported in arbitrary units, where a lower value indicates a higher/better muscle quality.
Body composition: skeletal muscle | Baseline
  CT scans will also be performed to assess skeletal muscle (SM). The L3 scan is uploaded into a software called SliceOmatic (TomoVision, Montreal, Quebec, Canada) to segment L3 into cross-sectional SM area, SAT area, and VAT area based on Hounsfield Units (HU) ranges: -29 to 150 for SM. An add-on module called Automated Body composition Analyzer using Computed tomography image Segmentation (ABACS) automatically performs the segmentation and produces an unbiased estimation.
Body composition: skeletal muscle | 12 weeks
  CT scans will also be performed to assess skeletal muscle (SM). The L3 scan is uploaded into a software called SliceOmatic (TomoVision, Montreal, Quebec, Canada) to segment L3 into cross-sectional SM area, SAT area, and VAT area based on Hounsfield Units (HU) ranges: -29 to 150 for SM. An add-on module called Automated Body composition Analyzer using Computed tomography image Segmentation (ABACS) automatically performs the segmentation and produces an unbiased estimation.
Body composition: skeletal muscle | 24 weeks
  CT scans will also be performed to assess skeletal muscle (SM). The L3 scan is uploaded into a software called SliceOmatic (TomoVision, Montreal, Quebec, Canada) to segment L3 into cross-sectional SM area, SAT area, and VAT area based on Hounsfield Units (HU) ranges: -29 to 150 for SM. An add-on module called Automated Body composition Analyzer using Computed tomography image Segmentation (ABACS) automatically performs the segmentation and produces an unbiased estimation.
Body composition: subcutaneous adipose tissue | Baseline
  CT scans will also be performed to subcutaneous adipose tissue (SAT). The L3 scan is uploaded into a software called SliceOmatic (TomoVision, Montreal, Quebec, Canada) to segment L3 into cross-sectional SM area, SAT area, and VAT area based on Hounsfield Units (HU) ranges: -190 to -30 for SAT. An add-on module called Automated Body composition Analyzer using Computed tomography image Segmentation (ABACS) automatically performs the segmentation and produces an unbiased estimation.
Body composition: subcutaneous adipose tissue | 12 weeks
  CT scans will also be performed to subcutaneous adipose tissue (SAT). The L3 scan is uploaded into a software called SliceOmatic (TomoVision, Montreal, Quebec, Canada) to segment L3 into cross-sectional SM area, SAT area, and VAT area based on Hounsfield Units (HU) ranges: -190 to -30 for SAT. An add-on module called Automated Body composition Analyzer using Computed tomography image Segmentation (ABACS) automatically performs the segmentation and produces an unbiased estimation.
Body composition: subcutaneous adipose tissue | 24 weeks
  CT scans will also be performed to subcutaneous adipose tissue (SAT). The L3 scan is uploaded into a software called SliceOmatic (TomoVision, Montreal, Quebec, Canada) to segment L3 into cross-sectional SM area, SAT area, and VAT area based on Hounsfield Units (HU) ranges: -190 to -30 for SAT. An add-on module called Automated Body composition Analyzer using Computed tomography image Segmentation (ABACS) automatically performs the segmentation and produces an unbiased estimation.
Body composition: visceral adipose tissue | Baseline
  CT scans will also be performed to assess visceral adipose tissue (VAT). The L3 scan is uploaded into a software called SliceOmatic (TomoVision, Montreal, Quebec, Canada) to segment L3 into cross-sectional SM area, SAT area, and VAT area based on Hounsfield Units (HU) ranges: -150 to -50 for VAT. An add-on module called Automated Body composition Analyzer using Computed tomography image Segmentation (ABACS) automatically performs the segmentation and produces an unbiased estimation.
Body composition: visceral adipose tissue | 12 weeks
  CT scans will also be performed to assess visceral adipose tissue (VAT). The L3 scan is uploaded into a software called SliceOmatic (TomoVision, Montreal, Quebec, Canada) to segment L3 into cross-sectional SM area, SAT area, and VAT area based on Hounsfield Units (HU) ranges: -150 to -50 for VAT. An add-on module called Automated Body composition Analyzer using Computed tomography image Segmentation (ABACS) automatically performs the segmentation and produces an unbiased estimation.
Body composition: visceral adipose tissue | 24 weeks
  CT scans will also be performed to assess visceral adipose tissue (VAT). The L3 scan is uploaded into a software called SliceOmatic (TomoVision, Montreal, Quebec, Canada) to segment L3 into cross-sectional SM area, SAT area, and VAT area based on Hounsfield Units (HU) ranges: -150 to -50 for VAT. An add-on module called Automated Body composition Analyzer using Computed tomography image Segmentation (ABACS) automatically performs the segmentation and produces an unbiased estimation.
Grip Strength | Baseline
  Grip strength will be assessed using a handgrip dynamometer. Grip strength is based on the maximal voluntary contraction of the subject's upper body muscles. One practice repetition is performed on each side. Three trials are performed on each side, alternating sides after every repetition. The maximal grip score from all six trials is recorded.
Grip Strength | 12 weeks
  Grip strength will be assessed using a handgrip dynamometer. Grip strength is based on the maximal voluntary contraction of the subject's upper body muscles. One practice repetition is performed on each side. Three trials are performed on each side, alternating sides after every repetition. The maximal grip score from all six trials is recorded.
Grip Strength | 24 weeks
  Grip strength will be assessed using a handgrip dynamometer. Grip strength is based on the maximal voluntary contraction of the subject's upper body muscles. One practice repetition is performed on each side. Three trials are performed on each side, alternating sides after every repetition. The maximal grip score from all six trials is recorded.
Muscle Power | Baseline
  Muscular power will be assessed using a linear position transducer (LPT). A sit-to-stand (STS) power test will be performed. Two practice repetitions are performed. Subsequently, three trial repetitions are performed, each with 60 seconds of rest in between. The greatest peak and mean power output in watts (W) of the three trial repetitions are used for analysis.
Muscle Power | 12 weeks
  Muscular power will be assessed using a linear position transducer (LPT). A sit-to-stand (STS) power test will be performed. Two practice repetitions are performed. Subsequently, three trial repetitions are performed, each with 60 seconds of rest in between. The greatest peak and mean power output in watts (W) of the three trial repetitions are used for analysis.
Muscle Power | 24 weeks
  Muscular power will be assessed using a linear position transducer (LPT). A sit-to-stand (STS) power test will be performed. Two practice repetitions are performed. Subsequently, three trial repetitions are performed, each with 60 seconds of rest in between. The greatest peak and mean power output in watts (W) of the three trial repetitions are used for analysis.
Fatigue: FACIT-F | Baseline
  Fatigue will be measured using the Functional Assessment of Chronic Illness Therapy Fatigue, a 1-page form that uses a rating scale that goes from 0 (no fatigue) to 10 (severe fatigue). It assesses the patient's fatigue levels in the last 7 days. It also measures how usual activities, performing work, walking, relationship, and enjoyment of life are affected by fatigue. A higher score indicates higher levels of perceived fatigue. Clinically meaningful changes are 3 points.
Fatigue: FACIT-F | 12 weeks
  Fatigue will be measured using the Functional Assessment of Chronic Illness Therapy Fatigue, a 1-page form that uses a rating scale that goes from 0 (no fatigue) to 10 (severe fatigue). It assesses the patient's fatigue levels in the last 7 days. It also measures how usual activities, performing work, walking, relationship, and enjoyment of life are affected by fatigue. A higher score indicates higher levels of perceived fatigue. Clinically meaningful changes are 3 points.
Fatigue: FACIT-F | 24 weeks
  Fatigue will be measured using the Functional Assessment of Chronic Illness Therapy Fatigue, a 1-page form that uses a rating scale that goes from 0 (no fatigue) to 10 (severe fatigue). It assesses the patient's fatigue levels in the last 7 days. It also measures how usual activities, performing work, walking, relationship, and enjoyment of life are affected by fatigue. A higher score indicates higher levels of perceived fatigue. Clinically meaningful changes are 3 points.
Depression and Anxiety | Baseline
  Depression will be measured using the Hospital Anxiety and Depression Scale (HADS), a concise, self-administered 1 page form that categorizes anxiety and depression. The total score goes from 0-21, and scores are categorized from minimal to severe depression/anxiety, with higher total scores indicate worse outcomes.
Depression and Anxiety | 12 weeks
  Depression will be measured using the Hospital Anxiety and Depression Scale (HADS), a concise, self-administered 1 page form that categorizes anxiety and depression. The total score goes from 0-21, and scores are categorized from minimal to severe depression/anxiety, with higher total scores indicate worse outcomes.
Depression and Anxiety | 24 weeks
  Depression will be measured using the Hospital Anxiety and Depression Scale (HADS), a concise, self-administered 1 page form that categorizes anxiety and depression. The total score goes from 0-21, and scores are categorized from minimal to severe depression/anxiety, with higher total scores indicate worse outcomes.
Bone Pain: FACT-BP | Baseline
  Bone pain will be determined using the FACT-BP questionnaire. FACT-BP is a 15-item scale assessing cancer-related bone pain and its effects on quality of life (QoL); the higher the aggregate score, the less the bone pain and/or the better the QoL. All scales score from 0-4 and a high scale score represents a higher response level. Minimal important differences for FACT-BP range from 3-7 points.
Bone Pain: FACT-BP | 12 weeks
  Bone pain will be determined using the FACT-BP questionnaire. FACT-BP is a 15-item scale assessing cancer-related bone pain and its effects on quality of life (QoL); the higher the aggregate score, the less the bone pain and/or the better the QoL. All scales score from 0-4 and a high scale score represents a higher response level. Minimal important differences for FACT-BP range from 3-7 points.
Bone Pain: FACT-BP | 24 weeks
  Bone pain will be determined using the FACT-BP questionnaire. FACT-BP is a 15-item scale assessing cancer-related bone pain and its effects on quality of life (QoL); the higher the aggregate score, the less the bone pain and/or the better the QoL. All scales score from 0-4 and a high scale score represents a higher response level. Minimal important differences for FACT-BP range from 3-7 points.
Quality of Life: FACT-P | Baseline
  Quality of life (QoL) will be measured using the Functional Assessment of Cancer Therapy-Prostate (FACT-P). The FACT-P is composed of both multi-item scales and single-item measures. These include physical, social, emotional, and functional well-being, along with an assessment of prostate-specific health status. five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All scales score from 0-4 and a higher score represents higher QoL. Clinically meaningful changes are 6-10 points.
Quality of Life: FACT-P | 12 weeks
  Quality of life (QoL) will be measured using the Functional Assessment of Cancer Therapy-Prostate (FACT-P). The FACT-P is composed of both multi-item scales and single-item measures. These include physical, social, emotional, and functional well-being, along with an assessment of prostate-specific health status. five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All scales score from 0-4 and a higher score represents higher QoL. Clinically meaningful changes are 6-10 points.
Quality of Life: FACT-P | 24 weeks
  Quality of life (QoL) will be measured using the Functional Assessment of Cancer Therapy-Prostate (FACT-P). The FACT-P is composed of both multi-item scales and single-item measures. These include physical, social, emotional, and functional well-being, along with an assessment of prostate-specific health status. five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All scales score from 0-4 and a higher score represents higher QoL. Clinically meaningful changes are 6-10 points.
Balance: NeuroCom | Baseline
  Balance will be assessed using the NeuroCom Smart Balance Master. A sensory organization test will be performed. An overall composite equilibrium score describing a person's overall level of performance during all of the trials in the sensory organization test is calculated, with a value between 0 and 100, with 0 indicating a large sway and loss of balance, and 100 indicating greater postural control. The composite score is a weighted-average of the following 14 scores: the condition 1 average score, the condition 2 average score, and the three equilibrium scores from each of the trials in conditions 3-6.
Balance: NeuroCom | 12 weeks
  Balance will be assessed using the NeuroCom Smart Balance Master. A sensory organization test will be performed. An overall composite equilibrium score describing a person's overall level of performance during all of the trials in the sensory organization test is calculated, with a value between 0 and 100, with 0 indicating a large sway and loss of balance, and 100 indicating greater postural control. The composite score is a weighted-average of the following 14 scores: the condition 1 average score, the condition 2 average score, and the three equilibrium scores from each of the trials in conditions 3-6.
Balance: NeuroCom | 24 weeks
  Balance will be assessed using the NeuroCom Smart Balance Master. A sensory organization test will be performed. An overall composite equilibrium score describing a person's overall level of performance during all of the trials in the sensory organization test is calculated, with a value between 0 and 100, with 0 indicating a large sway and loss of balance, and 100 indicating greater postural control. The composite score is a weighted-average of the following 14 scores: the condition 1 average score, the condition 2 average score, and the three equilibrium scores from each of the trials in conditions 3-6.
Arterial Stiffness: SphygmoCor | Baseline
  Arterial stiffness will be measured using the SphygmoCor Xcel (AtCor Medical). Arterial stiffness will be assessed using brachial pulse wave analysis (PWA) augmentation index and carotid-femoral pulse wave analysis (PWV). Greater PWA augmentation index and carotid-femoral PWV time indicates greater arterial stiffness, a surrogate end-point for cardiovascular disease.
Arterial Stiffness: SphygmoCor | 12 weeks
  Arterial stiffness will be measured using the SphygmoCor Xcel (AtCor Medical). Arterial stiffness will be assessed using brachial pulse wave analysis (PWA) augmentation index and carotid-femoral pulse wave analysis (PWV). Greater PWA augmentation index and carotid-femoral PWV time indicates greater arterial stiffness, a surrogate end-point for cardiovascular disease.
Arterial Stiffness: SphygmoCor | 24 weeks
  Arterial stiffness will be measured using the SphygmoCor Xcel (AtCor Medical). Arterial stiffness will be assessed using brachial pulse wave analysis (PWA) augmentation index and carotid-femoral pulse wave analysis (PWV). Greater PWA augmentation index and carotid-femoral PWV time indicates greater arterial stiffness, a surrogate end-point for cardiovascular disease.

OTHER OUTCOMES:
Self-Reported Physical Activity Levels | Baseline
  Physical activity levels will be determined using the Godin Leisure-Time Exercise questionnaire, a 1-page form that categorizes the number of minimal, moderate, and strenuous bouts of exercise lasting more than 15 minutes. Higher scores represent higher activity levels.
Self-Reported Physical Activity Levels | 12 weeks
  Physical activity levels will be determined using the Godin Leisure-Time Exercise questionnaire, a 1-page form that categorizes the number of minimal, moderate, and strenuous bouts of exercise lasting more than 15 minutes. Higher scores represent higher activity levels.
Self-Reported Physical Activity Levels | 24 weeks
  Physical activity levels will be determined using the Godin Leisure-Time Exercise questionnaire, a 1-page form that categorizes the number of minimal, moderate, and strenuous bouts of exercise lasting more than 15 minutes. Higher scores represent higher activity levels.
Physical Activity: accelerometry | Baseline
  Physical Activity will be quantified using accelerometers that will be worn continuously for ~1 wk after each visit to quantify sedentary, low, medium and high levels of activity.
Physical Activity: accelerometry | 12 weeks
  Physical Activity will be quantified using accelerometers that will be worn continuously for ~1 wk after each visit to quantify sedentary, low, medium and high levels of activity.
Physical Activity: accelerometry | 24 weeks
  Physical Activity will be quantified using accelerometers that will be worn continuously for ~1 wk after each visit to quantify sedentary, low, medium and high levels of activity.

CONTACTS AND LOCATIONS:
Overall Officials: Erik D Hanson, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The University of North Carolina will be adding and storing data on a secure, centralized server. No individual data will be made available to protect the identity of the patients in the trial.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials